CLINICAL TRIAL: NCT01768819
Title: The Effects of an Elderly-specific Multimodal Physical Activity Program: a Controlled Clinical Trial
Brief Title: Multimodal Physical Activity for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, José Rubens Rebelatto, Professor/Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01 - REVITA
Record Dates: First submitted 2013-01-12; First posted 2013-01-15 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Aging; Physical Activity
Keywords: aging; exercise; muscle strength; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Physical Activity
  Interventions: Behavioral: Physical Activity
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Physical Activity — The intervention consisted of elderly-specific physical activity program for one year. During this period a total of 123 physical activity sessions were carried out. Each session lasted 50 minutes and included stretching, aerobic endurance exercises, resistance exercises, activities involving coordination, agility and flexibility, respiratory exercises and relaxation exercises. The sessions took place three times a week, according to American College of Sports Medicine (ACSM) recommendations. Workloads were adjusted for each subject bimonthly according to their capacity. The sessions were standardized and carried out by previously trained physical educators.
  Arms: Intervention Group

SUMMARY:
Although some authors have observed favorable effects of group physical activity programs, others have reported that the individualized prescription of exercises may be jeopardized by programs that do not allow sufficient consideration of individual characteristics. Therefore, we aim to verify the effects of an elderly-specific multimodal physical activity program on physical parameters after one year of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the Geriatric Revitalization Program for one year
* Be on the waiting list for the Geriatric Revitalization Program

Exclusion Criteria:

* Attend less than 75% of the physical activity program's activities
* Absent any of the three follow-up physical parameter evaluations

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Static Balance | one year
  The one-leg stance test (OLST) was used to evaluate static balance. A point was marked at eye level on a board approximately one meter from the volunteer. Focusing on this point, the volunteer, with arms akimbo, lifted the leg of his or her choice by flexing the knee. The performance was timed with a chronometer (precision: 1ms) until either the individual lost balance or 30s was reached. The test was then carried out with the opposite leg and the series was repeated until three trials per leg had been performed. The mean time of the three trials was used for analysis.

SECONDARY OUTCOMES:
Aerobic Endurance | one year
  Aerobic endurance was measured using the one-mile test or the Rockport Walking Test, which consists of having subjects walk 1,609 meters quickly, but without running. The time spent performing the task and the final heart rate were measured.
Dynamic Balance | one year
  A maximum-speed walking test (MSWT) was used to measure dynamic balance. A course 3.33 m long and 33.3 cm wide was marked on the floor with tape and, beginning from a standing position, the participant walked the entire course as fast as possible without running when the signal was given. Three trials were carried out; the chronometer (precision: 1ms) was started as soon as the subject's foot crossed the starting line. The mean time from the trials was used for analysis.
Flexibility | one year
  A sit-and-reach test (SRT) with a modified Wells flexometer (precision: 1mm) was used to evaluate the flexibility of the trunk and upper limbs. The subjects sat on the floor with their soles flush against the lower edge of the device. Then, with their overlapped hands on the upper surface touching a sliding position marker, they pushed it forward along the scale while exhaling. The best of three trials was considered the result.
Handgrip Strength | one year
  Handgrip Strength was measured with a Jamar® hydraulic hand dynamometer (Sammons Preston Roylan, Bolingbrook, IL, USA) featuring a grading scale of 0-100 Kgf (precision: 2 Kgf). The best of three trials with the dominant upper limb was selected for analysis.
Body Mass Index | one year
  The weight and height were measured with a calibrated analogue scale with a stadiometer. The variable of weight was measured three times and the mean value considered. Such variables were used to calculate the BMI of the volunteers.
Body weight | one year
  The weight was measured with a calibrated analogue scale with a stadiometer. The variable was measured three times and the mean value considered.

CONTACTS AND LOCATIONS:
Overall Officials: José Rubens Rebelatto, Principal Investigator — Universidade Federal de Sao Carlos; Francisco Albuquerque-Sendín, Study Director — Universidade de Salamanca; Alessandra Paiva Castro, Study Chair — Universidade Federal do Espírito Santo; Thais Rabiatti Aurichio, Study Chair — Universidade Federal de Sao Carlos; Karla Helena Coelho Vilaça, Study Chair — Universidade Católica de Brasília; Victor da Silva Aquino, Study Chair — Universidade Federal de Sao Carlos